CLINICAL TRIAL: NCT00285051
Title: Study to Compare the Safety and Efficacy of 2 Different Doses of Inhaled D8-THC to Standard Therapy With Ondansetron in the Prevention of Acute Nausea From Moderately Emetogenic Chemotherapy
Brief Title: Comparison of Delta-8-THC to Ondansetron in the Prevention of Acute Nausea From Moderately Emetogenic Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug expiry date not extended
Sponsor: Rafa Laboratories (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Rafa protocol THC002/NVP
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: emesis, nausea,
MeSH Terms: conditions — Neoplasms; Vomiting; Nausea | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: Group 1 cycle 1 - Ondansetron; cycle 2 - 300 mcg of delta-8-THC per dose Group 2 cycle 1 - Ondansetron; cycle 2 - 600 mcg of delta-8-THC per dose Group 3 cycle 1 - 300 mcg of delta-8-THC per dose cycle 2 - Ondansetron Group 4 cycle 1 - 600 mcg of delta-8-THC per dose cycle 2 - Ondansetron
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Group 1 (Experimental): Chemo cycle 1 - IV Ondansetron Chemo cycle 2 - 300 mcg of delta-8-THC per dose
  Interventions: Drug: inhaled delta-8-THC 300mcg or 600mcg per dose
- Group 2 (Experimental): Chemo cycle 1 - IV Ondansetron Chemo cycle 2 - 600 mcg of delta-8-THC per dose
  Interventions: Drug: inhaled delta-8-THC 300mcg or 600mcg per dose
- Group 3 (Experimental): Chemo cycle 1 - 300 mcg of delta-8-THC per dose, Chemo cycle 2 - IV Ondansetron
  Interventions: Drug: inhaled delta-8-THC 300mcg or 600mcg per dose
- Group 4 (Experimental): Chemo cycle 1 - 600 mcg of delta-8-THC per dose Chemo cycle 2 - IV Ondansetron
  Interventions: Drug: inhaled delta-8-THC 300mcg or 600mcg per dose

INTERVENTIONS:
Drug: inhaled delta-8-THC 300mcg or 600mcg per dose — drugs to be used to prevent/treat nausea and/or vomiting due to cancer chemotherapy drug Patients will receive chemotherapy on day 0 and receive study medication, return on day 1or 2 and again on day 4 to return medication. There will be at least 10 days between the last dose of study medication from the first cycle and the first dose for the 2nd cycle..
  Patients will receive for each chemotherapy cycle either IV Ondansetron and Placebo inhalation, or IV Placebo and delta-8-THC inhalation. The patients will be randomized to receive one of 2 doses of the THC, either 300mcg or THC or 600mcg of THC
  Other Names: IV Ondansetron (comparator)

SUMMARY:
Patients will be treated for 2 consecutive chemo cycles with the study drug for one and placebo for the other. In addition, patients will receive an injection before the chemo, either ondansetron (if receiving placebo inhalation) or normal saline) if receiving active study drug. They will take study medication for 3 days, 4 times daily and fill out VAS scores before and after doses. Patients will be given rescue medication with each dose.

DETAILED DESCRIPTION:
The study is comparing the use of inhaled delata-8-THC in the prevention of nausea and vomitting in patients being treated with moderately emetogenic chemotherapy, and the patients will continue use for 3 days afterward. Patients will be given rescue medication and will fill out VAS scales for nausea, pain, appetite and dizziness. Patients will be treated for 2 cycles, one cycle receiving active drug (one of 2 doses) and the other placebo. Patients receiving placebo will receive ondansetron injection before chemo and patients receiving active drug will receive a normal saline injection. Patients will take the drug 4 times daily for 3 days. The patients will return to clinic for a visit after 24-48 hours and 4 days. Patients will bring a urine sample to measure metabolite. Patients will be given a diary to monitor dosing and side effects as well as concomitant medication. The study will be conducted in 2 - 3 centers. There will be 108 patients enrolled with 27 in each of 4 groups:

Group 1 cycle 1 - Placebo cycle 2 - 300 mcg of delta-8-THC per dose Group 2 cycle 1 - Placebo cycle 2 - 600 mcg of delta-8-THC per dose Group 3 cycle 1 - 300 mcg of delta-8-THC per doseGroup cycle 2 - Placebo Group 4 cycle 1 - 600 mcg of delta-8-THC per dose cycle 2 - placebo

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Man or woman between 18 and 85 years of age
* Patients who will be receiving at least 2 more cycles of moderately emetogenic chemotherapy
* Patients who are cognitively intact
* Performance Status of 60% or greater on the Karnofsky Scale
* Negative pregnancy test at screening visit in females of childbearing potential
* Use of appropriate contraceptive methods for females of childbearing potential during treatment (e.g. hormonal contraception, intrauterine device [IUD])

Exclusion Criteria:

* A history of psychiatric illness.
* A history of asthma and any other chronic respiratory illness.
* Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study.
* Serious illnesses such as asthma, diabetes mellitus, active peptic ulcer disease, infection, cardiovascular disease or any other disease which may affect the oucome parameters of this study
* Abnormal liver function tests (ALT, AST or AP > 2.5 x upper normal limit)
* Abnormal renal function (e.g. serum creatinine > 2 x upper normal limit)
* Abnormal pulmonary function test which in the judgment of the investigator is incompatible with inhalation of the study drug
* Known intolerance/hypersensitivity to study drugs (THC, ondansetron or dexamethasone) or drugs of similar chemical structure or pharmacological profile
* History of addiction to alcohol or drugs
* Existing or intended pregnancy or lactation
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
VAS scale for nausea | Up to 4 days after the patient receives chemotherapy. Measurements taken just before and 2 hours after inhalation morning and evening doses.
  subjective measurement of feeling of nausea. Patients to indicate on a horizontal line, how much nausea the patient feels, lower score = less nausea, higher score is more severe. Measurement is made on the line from "none" to "severe" for score.

SECONDARY OUTCOMES:
No. of emesis | up to the 4 days after patient receives chemotherapy
  number of times patient vomits recorded daily after receiving cancer chemotherapy
VAS scale for delayed nausea | Up to the 4 days after patient receives chemotherapy. Measurements taken just before and 2 hours after taking inhalation morning and evening doses. Delayed nausea is nausea that occurs 24 hours or more after receiving cancer chemotherapy.
  Subjective measurement of feeling of nausea. Patients to indicate on a horizontal line, lower score = less nausea, higher score is more severe. Measurement is made on the line from "none" to "severe" for score.
VAS scale for pain | Up to the 4 days after the patient takes the study medication after receiving chemotherapy. Measurements taken just before and 2 hours after inhalation morning and evening doses
  subjective measurement of feeling of pain at the moment Patients to indicate on a horizontal line, lower score = less pain, higher score is more severe pain. Measurement is made on the line from "none" to "severe" for score.
VAS scale for appetite stimulation | Up to 4 days after patient receives chemotherapy. Measurements are taken just before and 2 hours after taking inhalation morning and evening doses
  Patients to indicate on a horizontal line, lower score = less appetite, higher score is more appetite. Measurement is made on the line from "not at all" to "very hungry" for score.
VAS scale for dizziness | before and 2 hours after taking inhalation, morning and evening doses.
  subjective measurement of feeling dizzy Patients to indicate on a horizontal line, lower score = less nausea, higher score is more severe. Measurement is made on the line from "none" to "severe" for score.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Cherny, MD, Principal Investigator — Shaare Zedek Medical Center, Dept. of Oncology
Locations (2):
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Tel Litwinsky